CLINICAL TRIAL: NCT05033509
Title: Outcome of ECMO and CRRT, Experience of Hospital University MED VI, Oujda, Morocco.
Brief Title: Outcome of ECMO and CRRT.
Status: Completed | Type: Observational
Sponsor: Mohammed VI University Hospital (Other)
Responsible Party: Principal Investigator, Younes Oujidi, Principal Investigator, Mohammed VI University Hospital
Other Study IDs: Unite care
Record Dates: First submitted 2021-08-24; First posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Incidence of CRRT With ECMO Therapy; Mortality; and Renal Recovery
Keywords: COVID; AKI; CRRT; Ecmo

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ECMO and AKI
  Interventions: Other: supervision the Kidney fonction on ECMO

INTERVENTIONS:
Other: supervision the Kidney fonction on ECMO — patients who benefited from ECMO, and presented an acute kidney injury afterwards

SUMMARY:
Background:

Although acute kidney injury (AKI) is a frequent complication in patients receiving extracorporeal membrane oxygenation (ECMO), and the CRRT impact is widely studied. The incidence of simultaneous use of ECMO and CRRT remain unclear.

Objective: The investigatore conducted this retrospective study to define the incidence of concomitant CRRT with ECMO therapy and to determine the overall impact of this strategy on patient outcomes such as mortality and renal recovery.

Methods:

The investigatore retrospectively analyzed data of patients of all ages, genders and ethnicities, admitted in the intensive care unit of Mohammed VI University Hospital, Oujda, Morocco, on a cumulative period of 2 years (January 2019 - December 2020). Were enrolled in the study patients who benefited from ECMO, and presented an acute kidney injury afterwards, using 'Microsoft Excel' as a software to utilize the information collected from the computerized patient database. 30 patients were included in the final study.

ELIGIBILITY:
Inclusion Criteria:

* benefited from ECMO .
* presented an acute kidney injury afterwards

Exclusion Criteria:

* patients who developed AKI before benefitting from ECMO and/or missing data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We retrospectively analyzed data of patients of all ages, genders and ethnicities, admitted in the intensive care unit of Mohammed VI University Hospital, Oujda, Morocco, on a cumulative period of 2 years
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Ecmo and severe AKI requiring CRRT | through study completion, an average of 24 mounths
  2 groups of patient was identified on this study : first ones are how developped aki and needek CRRT , 2nd are those who developped aki without CRRT

CONTACTS AND LOCATIONS:
Locations (1):
- younes Oujidi, Berkane, Morocco

IPD SHARING:
Plan to Share IPD: No